CLINICAL TRIAL: NCT06473519
Title: A PHASE 3, RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE FORMULATED IN MULTIDOSE VIALS IN HEALTHY FEMALE ADULTS
Brief Title: A Study to Assess Safety, Tolerability and Immunogenicity of RSVpreF From Multidose Vials in Healthy Female Adults.
Acronym: Amélie
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C4841001; NCT06473519 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-06-17; First posted 2024-06-25 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: RSV infection; Multidose Vial (MDV); Single-dose Vial (SDV); 2-Phenoxyethanol (2-PE); Vaccines
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSVpreF multidose vial (MDV) (Experimental): RSVpreF with 2-PE formulated in an MDV
  Interventions: Biological: RSVpreF MDV
- RSVpreF single-dose vial (SDV) (Experimental): RSVpreF without 2-PE formulated in an SDV
  Interventions: Biological: RSVpreF SDV

INTERVENTIONS:
Biological: RSVpreF MDV — RSVpreF with 2-PE formulated in an MDV
  Arms: RSVpreF multidose vial (MDV)
Biological: RSVpreF SDV — RSVpreF without 2-PE formulated in an SDV
  Arms: RSVpreF single-dose vial (SDV)

SUMMARY:
Respiratory Syncytial Virus (RSV) is a common type of virus (germ) that can cause severe illness, where medical help is needed. RSV can lead to airway diseases in all ages. Vaccines help your body make antibodies. These antibodies help fight against diseases. This is called an immune response.

The purpose of this study is to learn about the safety, tolerability, and immunogenicity of a RSV vaccine called RSVpreF. RSVpreF comes either as:

* a single dose in a container (called a vial),
* or in a vial that holds multiple doses. A multidose vial contains more than one dose of RSVpreF.

  2-Phenoxyethanol (2-PE) is a preservative to help prevent the growth of bacteria (germs). This study will compare RSVpreF with an added preservative called 2-phenoxyethanol (2-PE) from a multidose vial, to RSVpreF without an added preservative, from a single-dose vial.

This study is looking to enroll nonpregnant, nonbreastfeeding, healthy female participants.

Participants will need to visit the study clinic two times during the study. Participants will also have a final safety telephone call at the end of the study. All participants will receive a single shot of the study vaccine either from:

* a multidose vial (with the preservative), or
* from a single-dose vial (without the preservative) at the first study clinic visit.

Blood samples will be taken at the two study clinic visits. Each participant will take part in the study for around 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy nonpregnant, nonbreastfeeding females 18 through 49 years of age at Visit 1 (Day 1).
2. Willing and able to comply with all scheduled visits, investigational plan, lifestyle considerations, and other study procedures.
3. Available for the duration of the study and can be contacted by telephone during study participation.
4. Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the ICD and in the protocol.

Exclusion Criteria:

1. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the vaccines being administered in the study.
3. Immunocompromised participants with known or suspected immunodeficiency, as determined by history, laboratory tests, and/or physical examination.
4. History or active autoimmune disease, including but not limited to systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin-dependent diabetes mellitus (type 1).
5. Bleeding diathesis or any condition that would, in the opinion of the investigator, contraindicate intramuscular injection.
6. Previous vaccination with any licensed or investigational RSV vaccine, or planned receipt of a nonstudy RSV vaccine throughout the study.
7. Receipt of chronic systemic treatment with immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before enrollment through conclusion of the study.
8. Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration or planned receipt throughout the study.
9. Current alcohol abuse or illicit drug use.
10. Individuals who are pregnant or breastfeeding.
11. Participation in other studies involving an investigational product within 28 days prior to study entry and/or during study participation. Participation in purely observational studies is acceptable.
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nonpregnant, nonbreastfeeding females
Enrollment: 453 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Qps-Mra, Llc, South Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Clinical Research Prime Rexburg, Rexburg, Idaho
  - Headlands Research - Detroit, Southfield, Michigan
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sarwar UN, Baker JB, Pereira L, Pahud BA, Finley J, Strong D, Pagnussat S, Patel S, Liu Y, Shittu E, Anastasiou OE, Kalinina EV, Swanson KA, Anderson AS, Gurtman A, Munjal I. Safety and immunogenicity of bivalent RSVpreF vaccine formulated in a multidose vial in healthy female participants in the USA: a multicentre, randomised, open-label, noninferiority phase 3 study. EClinicalMedicine. 2026 Jan 29;92:103767. doi: 10.1016/j.eclinm.2026.103767. eCollection 2026 Feb. PMID 41660362
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4841001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) either with the preservative formulated in a multiple dose vial (MDV) or without the preservative formulated in a single dose vial (SDV). Preservative used was 2-phenoxyethanol (2-PE).
Groups:
- RSVpreF (With Preservative, MDV): Participants were randomized to receive only a single 0.5 milliliter (mL) dose from MDV of RSVpreF (120 micrograms [mcg]), intramuscularly on Day 1.
- RSVpreF (Without Preservative, SDV): Participants were randomized to receive entire content from SDV of RSVpreF (120 mcg), intramuscularly on Day 1.
Period: Overall Study
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Started | 224 | 229
Vaccinated (on Day 1) | 223 | 227
Completed | 220 | 218
Not Completed | 4 | 11
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Randomized but not vaccinated | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all randomized participants who received study intervention.
Groups:
- RSVpreF (With Preservative, MDV): Participants were randomized to receive only a single 0.5 mL dose from MDV of RSVpreF (120 mcg), intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV) | Total
Number analyzed (Participants) | 223 | 227 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (9.3) | 34.4 (8.8) | 34.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 227 | 450
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 54 | 100
  Not Hispanic or Latino | 174 | 168 | 342
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 55 | 63 | 118
  White | 161 | 152 | 313
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Serum Neutralizing Titers (NTs) for Respiratory Syncytial Virus Subgroup A (RSV A) and Respiratory Syncytial Virus Subgroup B (RSV B) Before Vaccination
Description: GMTs and corresponding 2-sided 95% confidence intervals (CIs) were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution).
Time Frame: Before vaccination on Day 1
Population: Evaluable immunogenicity population (EIP): all eligible participants who received the study intervention to which they were randomized, had blood drawn for assay testing within the specified time frame (27 to 42 days after vaccination) for 1 month after vaccination, had at least 1 valid and determinate assay result at the 1-month follow-up visit, and had no major protocol violations. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 218 | 216
Titer
  RSV A: number analyzed (Participants) | 218 | 215
  RSV A | 2362 [2118.7 to 2634.0] | 2472 [2226.2 to 2744.8]
  RSV B | 2926 [2637.1 to 3245.7] | 3172 [2866.2 to 3509.8]

2. Primary Outcome: GMT and Geometric Mean Ratio (GMR) of Serum NTs for RSV A and RSV B at 1 Month After Vaccination
Description: GMTs and corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV A and B were reported in the descriptive data section of this outcome measure. GMR each for RSV A and RSV B was calculated as ratio of NTs of RSVpreF (MDV) to RSVpreF (SDV) and was reported in the statistical analysis section of this outcome measure.
Time Frame: 1 month after Vaccination on Day 1
Population: EIP: all eligible participants who received the study intervention to which they were randomized, had blood drawn for assay testing within the specified time frame (27 to 42 days after vaccination) for 1 month after vaccination, had at least 1 valid and determinate assay result at the 1-month follow-up visit, and had no major protocol violations. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 218 | 215
Titer
  RSV A | 33715 [30737.7 to 36981.4] | 35131 [31949.4 to 38630.0]
  RSV B | 41471 [37505.0 to 45856.0] | 45374 [40664.0 to 50628.8]
Statistical Analysis 1: Comparison: RSVpreF (With Preservative, MDV) vs RSVpreF (Without Preservative, SDV); RSV A; Test type: Non-Inferiority — Noninferiority of immune responses induced by MDVRSV preF compared to SDVRSV preF, assessed for RSVA&B at 1month after vaccination. Null hypotheses(H0): RSVA(H0A)=ln(μMDV)-ln(μSDV)<=-ln(1.5);RSVB(H0B):ln(μMDV)-ln(μSDV)<=-ln(1.5), where ln(μMDV)&ln(μSDV) are means of natural log-transformed antibody concentrations 1month after vaccination for MDV and SDV groups, respectively. Noninferiority=if lower bounds of 2-sided95%CI for GMT ratios (MDV/SDV) were >0.67(noninferiority margin=1.5)for RSVA&B; Geometric mean ratio = 0.96, 95% CI 2-sided [0.84 to 1.10] — GMR was calculated as group mean difference of logarithmically transformed antibody levels, back transformed to original units
Statistical Analysis 2: Comparison: RSVpreF (With Preservative, MDV) vs RSVpreF (Without Preservative, SDV); RSV B; Test type: Non-Inferiority — Noninferiority of immune responses induced by MDVRSV preF compared to SDVRSV preF, assessed for RSVA&B at 1 month after vaccination. Null hypotheses(H0):RSVA(H0A)=ln(μMDV)-ln(μSDV)<=-ln(1.5);RSVB(H0B):ln(μMDV)-ln(μSDV)<=-ln(1.5), where ln(μMDV)&ln(μSDV) are means of natural log-transformed antibody concentrations 1 month after vaccination for MDV and SDV groups, respectively. Noninferiority=if lower bounds of 2-sided 95%CI for GMT ratios(MDV/SDV) were >0.67(noninferiority margin=1.5)for RSVA&B; Geometric mean ratio = 0.91, 95% CI 2-sided [0.79 to 1.06] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions included redness, swelling and pain at injection site, reported in the electronic diary (e-diary) and the participant-reported reactogenicity (PARREACT) case report form (CRF). Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit= 0.5 centimeter (cm) and graded as mild: >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, Grade 4: necrosis (redness and swelling) or exfoliative dermatitis (redness). Pain at injection site was graded as mild: did not interfere with activity, moderate: interfered with activity, severe: prevented daily activity, Grade 4: emergency room visit or hospitalization for severe pain at injection site.
Time Frame: Day 1 through Day 7 after Vaccination
Population: Safety population consisted of all randomized participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 223 | 227
Percentage of participants
  Redness: Any | 9.4 [5.9 to 14.0] | 15.9 [11.4 to 21.3]
  Redness: Mild | 5.8 [3.1 to 9.8] | 9.3 [5.8 to 13.8]
  Redness: Moderate | 2.2 [0.7 to 5.2] | 6.2 [3.4 to 10.1]
  Redness: Severe | 1.3 [0.3 to 3.9] | 0.4 [0.0 to 2.4]
  Redness: Grade 4 | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Swelling: Any | 13.9 [9.6 to 19.1] | 14.1 [9.8 to 19.3]
  Swelling: Mild | 8.1 [4.9 to 12.5] | 8.8 [5.5 to 13.3]
  Swelling: Moderate | 4.9 [2.5 to 8.7] | 4.8 [2.4 to 8.5]
  Swelling: Severe | 0.9 [0.1 to 3.2] | 0.4 [0.0 to 2.4]
  Swelling: Grade 4 | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Pain at injection site: Any | 46.6 [39.9 to 53.4] | 52.9 [46.1 to 59.5]
  Pain at injection site: Mild | 37.2 [30.9 to 43.9] | 43.6 [37.1 to 50.3]
  Pain at injection site: Moderate | 9.4 [5.9 to 14.0] | 8.4 [5.1 to 12.8]
  Pain at injection site: Severe | 0 [0.0 to 1.6] | 0.9 [0.1 to 3.1]
  Pain at injection site: Grade 4 | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]

4. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, vomiting, nausea, diarrhea, muscle pain and joint pain, recorded in the e-diary and PARREACT CRF. Fever measured in degree Celsius and ranged: mild (38.0 - 38.4); moderate (38.5 - 38.9); severe (39.0 - 40.0); Grade 4: >40.0. Fatigue, headache, nausea, muscle and joint pain graded as: mild (didn't interfere with activity); moderate (some interference with activity); severe (prevented daily routine activity); Grade 4 [emergency room (ER) visit or hospitalization). Vomiting graded as: mild (1-2 times in 24 hours[h]); moderate (>2 times in 24h); severe (required intravenous hydration); Grade 4 (ER visit or hospitalization). Diarrhea graded as: mild (2-3 loose stools in 24h); moderate (4-5 loose stools in 24h); severe (6 or more loose stools in 24h); Grade 4 (ER visit or hospitalization).
Time Frame: Day 1 through Day 7 after Vaccination
Population: Safety population consisted of all randomized participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 223 | 227
Percentage of participants
  Fever: Any | 3.1 [1.3 to 6.4] | 1.8 [0.5 to 4.5]
  Fever: Mild | 1.8 [0.5 to 4.6] | 0.9 [0.1 to 3.2]
  Fever: Moderate | 0.4 [0.0 to 2.5] | 0.4 [0.0 to 2.5]
  Fever: Severe | 0.9 [0.1 to 3.2] | 0.4 [0.0 to 2.5]
  Fever: Grade 4 | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Fatigue: Any | 47.5 [41.0 to 54.5] | 46.7 [40.4 to 53.9]
  Fatigue: Mild | 20.6 [15.6 to 26.7] | 21.1 [16.2 to 27.3]
  Fatigue: Moderate | 25.1 [19.7 to 31.5] | 24.7 [19.4 to 31.1]
  Fatigue: Severe | 1.8 [0.5 to 4.5] | 0.9 [0.1 to 3.2]
  Fatigue: Grade 4 | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Headache: Any | 36.8 [30.6 to 43.7] | 39.2 [33.1 to 46.3]
  Headache: Mild | 22.4 [17.2 to 28.6] | 22.9 [17.8 to 29.2]
  Headache: Moderate | 13.5 [9.3 to 18.7] | 15.4 [11.1 to 21.0]
  Headache: Severe | 0.9 [0.1 to 3.2] | 0.4 [0.0 to 2.5]
  Headache: Grade 4 | 0 [0.0 to 1.6] | 0.4 [0.0 to 2.5]
  Nausea: Any | 19.3 [14.4 to 25.2] | 15.4 [11.1 to 21.0]
  Nausea: Mild | 13.5 [9.3 to 18.7] | 11.0 [7.3 to 16.0]
  Nausea: Moderate | 4.9 [2.5 to 8.7] | 4.4 [2.2 to 8.0]
  Nausea: Severe | 0.4 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Nausea: Grade 4 | 0.4 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Muscle Pain: Any | 38.6 [32.3 to 45.5] | 31.7 [26.0 to 38.5]
  Muscle Pain: Mild | 25.1 [19.7 to 31.5] | 19.4 [14.6 to 25.3]
  Muscle Pain: Moderate | 13.0 [8.9 to 18.2] | 12.3 [8.4 to 17.5]
  Muscle Pain: Severe | 0.4 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Muscle Pain: Grade 4 | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Joint Pain: Any | 14.8 [10.5 to 20.2] | 19.4 [14.6 to 25.3]
  Joint Pain: Mild | 8.5 [5.2 to 13.0] | 11.9 [8.1 to 17.0]
  Joint Pain: Moderate | 6.3 [3.5 to 10.4] | 7.5 [4.5 to 11.8]
  Joint Pain: Severe | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Joint Pain: Grade 4 | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Vomiting: Any | 3.6 [1.6 to 7.0] | 2.2 [0.7 to 5.1]
  Vomiting: Mild | 3.1 [1.3 to 6.4] | 1.8 [0.5 to 4.5]
  Vomiting: Moderate | 0 [0.0 to 1.6] | 0.4 [0.0 to 2.5]
  Vomiting: Severe | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Vomiting: Grade 4 | 0.4 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Diarrhea: Any | 17.5 [12.8 to 23.2] | 18.1 [13.4 to 23.9]
  Diarrhea: Mild | 11.7 [7.8 to 16.7] | 15.0 [10.7 to 20.5]
  Diarrhea: Moderate | 4.9 [2.5 to 8.7] | 3.1 [1.3 to 6.3]
  Diarrhea: Severe | 0.4 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Diarrhea: Grade 4 | 0.4 [0.0 to 2.5] | 0 [0.0 to 1.6]

5. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention were included in evaluation of this outcome measure. AEs included both serious AEs (SAEs) and all non-SAEs. Events collected by systematic assessment (local reactions and systemic events) were excluded from evaluation.
Time Frame: Within 1 Month after Vaccination
Population: Safety population consisted of all randomized participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 223 | 227
Percentage of participants | 9.0 [5.6 to 13.5] | 8.4 [5.1 to 12.8]

6. Primary Outcome: Percentage of Participants With SAEs Throughout the Study
Description: An AEs was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and other important medical events per protocol of the study. Events collected by systematic assessment (local reactions and systemic events) were excluded from evaluation.
Time Frame: Within 42 to 49 days after Vaccination on Day 1 (maximum up to 1.6 months)
Population: Safety population consisted of all randomized participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 223 | 227
Percentage of participants | 0.4 [0.0 to 2.5] | 0.9 [0.1 to 3.1]

7. Secondary Outcome: Percentage of Participants Achieving Seroresponse for RSV A and RSV B of Serum NTs at 1 Month After Vaccination
Description: Seroresponse was defined as achieving a >=4-fold rise from baseline (before vaccination) if the baseline measurement was above the lower limit of quantification (LLOQ). If the baseline measurement was below the LLOQ, a postvaccination assay result >=4*LLOQ was considered a seroresponse.
Time Frame: 1 Month after Vaccination
Population: EIP was analyzed. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
Number analyzed (Participants) | 218 | 215
Percentage of participants
  RSV A: number analyzed (Participants) | 218 | 214
  RSV A | 91.7 [87.3 to 95.0] | 91.6 [87.0 to 94.9]
  RSV B | 96.8 [93.5 to 98.7] | 90.7 [86.0 to 94.2]

ADVERSE EVENTS:
Time Frame: Systematic assessment (local reactions and systemic events): Day 1 through Day 7 after Vaccination; Non-systematic assessment (serious AEs and all-cause mortality): within 42 to 49 days after Vaccination on Day 1 (maximum up to 1.6 months), Other AEs: within 1 month after Vaccination
Description: Same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population consisted of all randomized participants who received study intervention.
Arm/Group | RSVpreF (With Preservative, MDV) | RSVpreF (Without Preservative, SDV)
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/227
Serious Adverse Events (participants affected / at risk) | 1/223 | 2/227
Other Adverse Events (participants affected / at risk) | 169/223 | 174/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSVpreF (With Preservative, MDV) (N=223) | RSVpreF (Without Preservative, SDV) (N=227)
Anaphylactic reaction (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSVpreF (With Preservative, MDV) (N=223) | RSVpreF (Without Preservative, SDV) (N=227)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (FATIGUE) (General disorders) | 106 | 106
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 104 | 120
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (FEVER) (General disorders) | 7 | 4
Swelling (SWELLING) (General disorders) | 31 | 32
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 39 | 41
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Nausea (NAUSEA) (Gastrointestinal disorders) | 43 | 35
Vomiting (VOMITING) (Gastrointestinal disorders) | 8 | 5
Milk allergy (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Onychomycosis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 33 | 44
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 86 | 72
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain fog (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (HEADACHE) (Nervous system disorders) | 82 | 89
Hypoaesthesia (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 0 | 1
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 21 | 36
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT06473519/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT06473519/SAP_001.pdf